CLINICAL TRIAL: NCT06409312
Title: Assessing the Feasibility of a Digital Healthcare App for Patient Rehabilitation After Total Hip Arthroplasty
Brief Title: Digital Healthcare App After Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-D0008
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Akina Cloud (Experimental)
  Interventions: Device: Akina Cloud

INTERVENTIONS:
Device: Akina Cloud — Akina Cloud is a digital health application that supports the therapeutic training of people with musculoskeletal conditions. It provides two therapeutic training programs for patients, one for each specific indication. Patients have continuous access to these programs through Akina Cloud, allowing them to independently complete nine training sessions without supervision. A minimum of three sessions per week is recommended, but patients have the option to engage in daily sessions if preferred. These therapy programs are based on current treatment guidelines and supported by relevant scientific research. They include customizable physical exercises tailored to individual needs and difficulty levels. Patients receive audio-visual guidance during these exercise sessions to ensure proper execution. Exercise therapy has demonstrated its ability to reduce pain, improve physical function, and enhance the overall quality of life for patients suffering from back pain and hip osteoarthritis.

SUMMARY:
This study examines the effectiveness of rehabilitation after hip replacement surgery using a specialised app called Akina Cloud. Medical professionals at the Schulthess Clinic will provide detailed information about the study. Participants must meet certain eligibility requirements. There will be time for consideration before enrolment. A demonstration of how to use the app will be provided upon agreement. Participants will be shown how to set up their profile and interact with a real therapist who will provide feedback. The initial 30-minute introduction is scheduled to take place a few days after surgery while still in hospital. Participants will be asked to complete several questionnaires. The rehabilitation process involves using the app for at least 12 weeks, at least three times a week, for 20-30 minutes per session. Direct communication with the therapist via the app is available for any queries. Follow-up questionnaires will be emailed at 6 and 12 weeks, after training, and again at 26 weeks to assess progress and feedback on the use of the app. Each session with the app lasts about 20 minutes and the questionnaire takes about 30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Unilateral initial implantation of a minimally-invasive hip endoprosthesis
* Age between 18 and 75 years old
* Ownership of a private laptop or desktop computer
* Stable internet connection at home
* Familiarity with the use of laptop or desktop computer

Exclusion Criteria:

* Bilateral initial implantation of a minimally-invasive hip endoprosthesis
* Not fluent in German or English
* Other conditions where active therapy is contraindicated
* Neurological diseases that limit the ability to walk
* Chronic lower limb pain
* Rheumatological diseases
* Other inflammatory diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-21 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of completed training sessions and the number of repetitions per sessionweeks of training. | after 12 weeks

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) | Baseline, 6 weeks, 12 weeks
  Intrinsic motivation inventory (IMI) consists of 6 subscales, the items are rated on a Likert scale ranging from 1 ("not at all true") to ("very true") for each item. A higher score indicates stronger intrinsic motivation.
Net Promoter Score (NPS) | 6 weeks, 12 weeks
  The NPS is a metric used to assess customer loyalty and satisfaction by asking a single question: "How likely is it that you would recommend our company/product/service to a friend or colleague?"The scale ranges form 0 to 10. A higher score indicates stronger intrinsic motivation.
Post-Study System Usability Questionnaire (PSSUQ) | 6 weeks, 12 weeks
  The Post-Study System Usability Questionnaire is a standardised questionnaire desigend to evaluate users' perceptions of the usability of a system of product after they have interacted with it.The questionnaire consists of a set of Likert-scale questions that cover various aspects of the user experience. The lower the score, the better the performance and satisfaction.
Hip disability and Osteoarthritis Outcome Score | 6 weeks, 12 weeks, 26 weeks
  The Hip disability and Osteoarthritis Outcome Score is a self-report questionnnaire with five subsets (pain, symptoms, activities of daily living, sports and recreations and quality in life). The scores range from 0 to 100, where a higehr score indicate less ssymptoms and disability.
International Physical Activity Questionnaire | 6 weeks, 12 weeks, 26 weeks
  The questionnaire covers activities such as work-related, transportation, household chores, and leisure-time activities. The responses are then used to categorise individuals into different levels of physical activity, ranging from low to high.

IPD SHARING:
Plan to Share IPD: No